CLINICAL TRIAL: NCT07052084
Title: Systematic Adjunction of Vasopressine in Hyperkinetic Septic Shock Patients - A Multicentric RCT
Brief Title: Systematic Adjunction of Vasopressine in Septic Shock
Acronym: SAVSepticShock
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCAPHM23_0465; 2024-513401-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Septic Shock
Keywords: Vasopressine; Systematic adjunction
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vassopressine (Experimental)
  Interventions: Drug: Vasopressin administration
- Placebo (Placebo Comparator)
  Interventions: Drug: Sodium chloride administration

INTERVENTIONS:
Drug: Vasopressin administration — Low dose of vasopressin (0.02ui /min), maximum 5 days
  Arms: Vassopressine
Drug: Sodium chloride administration — NaCl 0.9 %, maximum 5 days
  Arms: Placebo

SUMMARY:
Septic shock is a syndrome associated with severe infection and a mortality rate of approximately 45%. In line with current recommendations, norepinephrine is the first-line vasopressor used in patients with septic shock. In a previous study, norepinephrine doses above 1 µg/kg/min were associated with mortality rates over 90%. In the same study, doses above 0.3 µg/kg/min were associated with a mortality rate of 40%. An increased mortality compared to the general 40% mortality of septic shock appears to be associated with norepinephrine doses as low as 0.3 µg/kg/min.

Vasopressin stimulates V1 receptors, primarily located on vascular smooth muscle cells. When V1a receptors are stimulated, they induce vasoconstriction by activating protein kinase C via a Gq protein and various second messengers.

Its use is validated in refractory shock states by international guidelines as a second-line vasopressor. This indication was further reinforced in the 2021 update of the septic shock management recommendations.

The VASST study, a randomized controlled trial, assessed the effects of vasopressin versus norepinephrine in septic shock. It found no overall difference in mortality between the two groups. However, in less severe cases where norepinephrine doses were below 14 µg/min before randomization, vasopressin was associated with significantly lower mortality, suggesting potential benefits from early introduction of a second vasopressor.

The VANISH trial failed to confirm this hypothesis, possibly due to broad inclusion criteria and unclear protocol regarding the combined use of both agents. Our hypothesis is that (1) vasopressin is beneficial when used synergistically with norepinephrine; (2) due to its negative effect on cardiac output (as shown in previous studies), vasopressin should only be administered to patients in the hyperdynamic phase of septic shock.

The hypothesis is that the systematic addition of vasopressin to norepinephrine therapy in a hyperdynamic septic shock subpopulation would improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Patient who has consented to take part in the research or patient whose close relative has consented to take part in the research or, failing that, patient being included in an emergency situation
* Patient in septic shock with adapted cardiac output
* Patient in whom noradrenaline dosage has been greater than 0.3μg/kg/min for less than 12 hours
* Patients benefiting from or affiliated to social security

Exclusion Criteria:

* Patient with acute coronary syndrome
* Patient with known history of acute coronary syndrome
* Patient with suspected mesenteric ischemia
* Patient with hyponatremia < 130mmol/L,
* Known allergy to vasopressin or its excipients
* Minors
* Pregnant women
* Patients under legal guardianship or curatorship
* Patients under judicial protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
SOFA score comparison between the two groups | 48 hours after administration of experimental drug (H48)
  Sepsis-related Organ Failure Assessment, 0 to 24 points (higher scores indicate more severe organ dysfunction)

SECONDARY OUTCOMES:
SOFA score comparison between the two groups | 120 hours after administration of experimental drug (H120)
  Sepsis-related Organ Failure Assessment, 0 to 24 points (higher scores indicate more severe organ dysfunction)
Mortality comparison between the two groups | 28 days after administration of experimental drug (D28)
Lactatemia decrease comparison between the two groups | Between administration of experimental drug (H0), 24 hours after (H24), and 48 hours after (H48)
Noradrenaline use comparison between the two groups | 5 days after administration of experimental drug (D5)
  Maximum dose
Renal function comparison between the two groups | 28 days after administration of experimental drug (D28)
  Number of days alive without renal replacement therapy
Respiratory function comparison between the two groups | 28 days after administration of experimental drug (D28)
  Number of days alive without mechanical ventilation
Occurrence of myocardial ischemia comparison between the two groups | 28 days after administration of experimental drug (D28)
Occurrence of cardiogenic shock comparison between the two groups | 28 days after administration of experimental drug (D28)
Occurrence of mesenteric ischemia comparison between the two groups | 28 days after administration of experimental drug (D28)
Occurrence of digital ischemia comparison between the two groups | 28 days after administration of experimental drug (D28)
Occurrence of atrial fibrillation comparison between the two groups | 28 days after administration of experimental drug (D28)
Occurrence of a thromboembolic event comparison between the two groups | 28 days after administration of experimental drug (D28)

CONTACTS AND LOCATIONS:
Overall Officials: François Crémieux, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No